CLINICAL TRIAL: NCT00909142
Title: Bonefos and the Consumption of Analgesics. Influence of Clodronate on Analgesics Consumption Among Patients With Bone Metastasis
Brief Title: Bonefos and the Consumption of Analgesics
Acronym: BICAM
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Healthcare AG
Other Study IDs: 14236; Bonefos
Record Dates: First submitted 2009-05-25; First posted 2009-05-27 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Bone Neoplasms
Keywords: Breast cancer; Prostate cancer; Multiple myeloma
MeSH Terms: conditions — Bone Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Multiple Myeloma | interventions — Clodronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group1
  Interventions: Drug: Bonefos (Clodronate, BAY94-8393)

INTERVENTIONS:
Drug: Bonefos (Clodronate, BAY94-8393) — Patients in regular clinical practice receiving Bonefos according to local drug information

SUMMARY:
The effect of Bonefos on consumption of analgesics (drugs used for pain treatment) in patients with proven bone metastases.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer or prostate cancer or multiple myeloma.
* Bone metastasis.
* Ability to use analgesics and clodronate 1600 mg/day.

Exclusion Criteria:

* Hypersensitivity to bisphosphonates.
* Clodronate in previous therapy.
* Concomitant use of other bisphosphonates.
* Serious renal insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Random sample of cancer patients visting oncologist or urologist ambulance who are suitable for standard clodronate treatment.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Analgesics consumption after 12 months of treatment with Bonefos in patients with bone metastases and breast or prostate cancer or multiple myeloma | 12 months

SECONDARY OUTCOMES:
Decrease in pain measured by VAS (Visual Analogue Scale) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Czechia